CLINICAL TRIAL: NCT04340440
Title: Surgical and Oncologic Outcomes After Curative D2 vs D1 Gastrectomy in Operable Gastric Carcinoma, A Randomized Controlled Study in Egyptian Population
Brief Title: Curative D2 vs D1 Lymphadenectomy in Operable Gastric Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mohamed El Messiry, Ass. Professor, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0302764
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Gastric Cancer
Keywords: Operable gastric cancer; D2 vs D1 lymphadenectomy; Surgical and Oncologic outcomes
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Randomization by opaque sealed envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D1 lymphadenectomy (Active Comparator): Operable gastric cancer was treated by radical gastrectomy and limited D1 lymphadenectomy
  Interventions: Procedure: D1 lymphadenectomy
- D2 lymphadenectomy (Active Comparator): Operable gastric cancer was treated by radical gastrectomy and extended D2 lymphadenectomy
  Interventions: Procedure: D2 lymphadenectomy

INTERVENTIONS:
Procedure: D1 lymphadenectomy — Radical gastrectomy with D1 lymphadenectomy
  Arms: D1 lymphadenectomy
Procedure: D2 lymphadenectomy — Radical gastrectomy with D2 lymphadenectomy
  Arms: D2 lymphadenectomy

SUMMARY:
Gastric carcinoma is the second most common cause of cancer-related deaths and its main treatment modality if potentially curable is surgery but the optimal surgical resection is controversial. The aim of the current study was to assess the outcomes of curative D2 compared to D1 gastrectomy of operable gastric carcinoma regarding postoperative morbidity and mortality, disease recurrence and survival rates.

DETAILED DESCRIPTION:
80 consecutive patients with potentially operable gastric carcinoma were randomized via concealed envelopes into 2 groups (each included 40 patients), group I managed by radical gastrectomy with D1 lymphadenectomy while group II managed by radical gastrectomy with D2 lymphadenectomy . Both groups were compared regarding postoperative mortality, morbidities, tumor recurrence and 2 years survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric carcinoma
* Potentially operable gastric carcinoma without evidence of distant metastasis

Exclusion Criteria:

* Complicated gastric cancer (obstructed or perforated)
* Locally irresectable tumor
* Previous or coexisting cancer
* Prior gastric surgery or neoadjuvant chemotherapy
* Contraindication for major surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Postoperative morbidity rate | 30 days after surgery
  Frequency of early postoperative complications
Operative mortality rate | Within 30 days after surgery
  Frequency of early postoperative mortality

SECONDARY OUTCOMES:
2 years Recurrence rate | 2 years after surgery
  Frequency of tumor recurrence within 2 years after curative surgery
2 years Cancer specific mortality rate | 2 years after surgery
  Frequency of patients died because of gastric cancer within 2 years after curative surgery
2 years Disease free survival rate | 2 years after surgery
  Percentage of patients survived for 2 years without tumor recurrence
2 years Overall survival rate | 2 years after surgery
  Percentage of patients survived for 2 years with/without tumor recurrence

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hartgrink HH, van de Velde CJ, Putter H, Bonenkamp JJ, Klein Kranenbarg E, Songun I, Welvaart K, van Krieken JH, Meijer S, Plukker JT, van Elk PJ, Obertop H, Gouma DJ, van Lanschot JJ, Taat CW, de Graaf PW, von Meyenfeldt MF, Tilanus H, Sasako M. Extended lymph node dissection for gastric cancer: who may benefit? Final results of the randomized Dutch gastric cancer group trial. J Clin Oncol. 2004 Jun 1;22(11):2069-77. doi: 10.1200/JCO.2004.08.026. Epub 2004 Apr 13. PMID 15082726
- [Background] Wu CW, Hsiung CA, Lo SS, Hsieh MC, Chen JH, Li AF, Lui WY, Whang-Peng J. Nodal dissection for patients with gastric cancer: a randomised controlled trial. Lancet Oncol. 2006 Apr;7(4):309-15. doi: 10.1016/S1470-2045(06)70623-4. PMID 16574546
- [Background] Tamura S, Takeno A, Miki H. Lymph node dissection in curative gastrectomy for advanced gastric cancer. Int J Surg Oncol. 2011;2011:748745. doi: 10.1155/2011/748745. Epub 2011 Jun 14. PMID 22312521